CLINICAL TRIAL: NCT06446596
Title: Effect of the Implementation of Telerehabilitation-based Exercises Compared to the Standard Use of Exercise Dossier and Intervention Diary in a Home Therapeutic Exercise Intervention in Patients With Low Back Pain
Brief Title: Telerehabilitation-based Exercises vs Standard Home-based Exercise in Low Back Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Rodrigo Martín-San-Agustin, Assistant Professor of Physiotherapy, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Telerehab_Low_back_pain
Record Dates: First submitted 2024-05-31; First posted 2024-06-06 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Low Back Pain
Keywords: low back pain; exercise; telerehabilitation
MeSH Terms: conditions — Low Back Pain; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Telerehabilitation-based exercises (Experimental): Home therapeutic exercise intervention scheduled through a software of digital physiotherapy and telerehabilitation
  Interventions: Other: Exercise supported by the digital physiotherapy and telerehabilitation software TRAK
- Standard home-based exercise (Active Comparator): Home therapeutic exercise program scheduled through a dossier and an exercise diary
  Interventions: Other: Standard home-based exercise

INTERVENTIONS:
Other: Exercise supported by the digital physiotherapy and telerehabilitation software TRAK — 8 week home therapeutic exercise program that includes flexibility and strength exercises scheduled through the software a digital physiotherapy and telerehabilitation. The program will be carried out with a frequency of 3 weekly sessions, preferably on alternate days. The program will be carried out with the support of the TRAK software (https://www.trakphysio.com/es/), which allows the exercises to be carried out in front of a camera that, with the help of an artificial intelligence system, offers feedback to the participant and allows you to keep a record of the sessions. As an addition to the home sessions, two face-to-face sessions will be held in the first and fifth weeks, respectively. The exercise program includes three levels of difficulty (easy, intermediate and difficult), with patients advancing to subsequent levels once each level is successfully overcome.
  Arms: Telerehabilitation-based exercises
Other: Standard home-based exercise — 8 week home therapeutic exercise program that includes flexibility and strength exercises scheduled through a dossier and an exercise diary. The program will be carried out with a frequency of 3 weekly sessions, preferably on alternate days. The program will be carried out with the support of an information dossier of the exercises to be performed and a monitoring diary in which everything related to the sessions carried out will be noted.. As an addition to the home sessions, two face-to-face sessions will be held in the first and fifth weeks, respectively. The exercise program includes three levels of difficulty (easy, intermediate and difficult), with patients advancing to subsequent levels once each level is successfully overcome.
  Arms: Standard home-based exercise

SUMMARY:
The objective of the study is to compare the effect of a telerehabilitation-based exercise program, versus a home therapeutic exercise program scheduled through a dossier and an exercise diary, with respect to disability (measured using the OSWESTRY questionnaire) and other variables (range of motion, strength, fatigue, histological changes, pain, medication intake, psychosocial factors and adherence), in patients with low back pain.

DETAILED DESCRIPTION:
The objective of the study is to compare the effect of a telerehabilitation-based exercise program, versus a home therapeutic exercise program scheduled through a dossier and an exercise diary, with respect to disability (measured using the OSWESTRY questionnaire) and other variables (range of motion, strength, fatigue, histological changes, pain, medication intake, psychosocial factors and adherence), in patients with low back pain.

This randomized controlled trial has a parallel design, with two groups. Both groups will complete an 8-week home exercise program that includes flexibility and strength exercises. The program will be carried out with a frequency of 3 weekly sessions, preferably on alternate days. In the case of the experimental group, the program will be carried out with the support of the TRAK computer tool (https://www.trakphysio.com/es/), which allows the exercises to be carried out in front of a camera that, with the help of an artificial intelligence system, offers feedback to the participant and allows investigators/clinicians to keep a record of the sessions. In the case of the control group, the program will be carried out with the support of an information dossier of the exercises to be performed and a monitoring diary in which everything related to the sessions carried out will be noted. In both groups, as an addition to the home sessions, two face-to-face sessions will be held in the first and fifth weeks, respectively.

The exercise program includes flexibility and strength exercises, each made up of three levels of difficulty (easy, intermediate and difficult), with patients advancing to subsequent levels once each level is successfully overcome.

ELIGIBILITY:
Inclusion Criteria:

* Nonspecific subacute or chronic low back pain

Exclusion Criteria:

* Neuropathic pain
* Pain below the knees
* Pain in legs with tingling, sensation of current or sensory alterations
* Positive neurological tests. Lack of strength, sensitivity or altered reflexes
* Canal stenosis
* Nociplastic pain (fibromyalgia, generalized pain, emotional lability, affective and cognitive implications)
* Previous lumbar surgery
* Specific pathology (rheumatic, spondylolisthesis, oncological, fractures...)
* Pregnancy
* Performing medium-high intensity exercise of more than 100 minutes a week
* Pathology that prevents exercise (decompensated cardiac pathology, decompensated respiratory pathology, significant mobility difficulties...)
* Lack of digital skills
* Visual problems that prevent exercise with the phone screen

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-11-04 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Disability | 8 weeks measurement (post intervention)
  Disability measured using the Oswestry Disability Index

SECONDARY OUTCOMES:
Disability | Baseline; 32 weeks measurement (24 weeks post intervention)
  Disability measured using the Oswestry Disability Index (range score from 0 [less disability] to 100 [more disability])
Range of movement (Schober score) | Baseline; 8 weeks measurement (post intervention); 32 weeks measurement (24 weeks post intervention)
  Range of movement measured using the modified Schober score (a higher score is an indicator of better range of movement)
Range of movement (Finger floor distance test) | Baseline; 8 weeks measurement (post intervention); 32 weeks measurement (24 weeks post intervention)
  Range of movement measured using the Finger floor distance test (a lower distance is an indicator of better range of movement)
Extensor low back muscle strength | Baseline; 8 weeks measurement (post intervention); 32 weeks measurement (24 weeks post intervention)
  Extensor low back muscle strength measured using the Biering-Sorensen test (a higher score is an indicator of better strength)
Muscle thickness (low back extensor muscles) | Baseline; 8 weeks measurement (post intervention); 32 weeks measurement (24 weeks post intervention)
  Muscle thickness (low back extensor muscles) measured using ultrasonography
Muscle thickness (transversus abdominis) | Baseline; 8 weeks measurement (post intervention); 32 weeks measurement (24 weeks post intervention)
  Muscle thickness (transversus abdominis) measured using ultrasonography
Low Back Pain | Baseline; 8 weeks measurement (post intervention); 32 weeks measurement (24 weeks post intervention)
  Mean pain during last week measured with a numerical pain rating scale (range score from 0 [no pain] -10 [worst pain])
Medication intake | Baseline; 8 weeks measurement (post intervention); 32 weeks measurement (24 weeks post intervention)
  Medication intake registered using a diary
Kinesiphobia | Baseline; 8 weeks measurement (post intervention); 32 weeks measurement (24 weeks post intervention)
  Kinesiofobia measured using the Tampa Scale of Kinesiofobia (range score from 17 [lower levels of kinesiophobia]-68 [higher levels of kinesiophobia])
Depression | Baseline; 8 weeks measurement (post intervention); 32 weeks measurement (24 weeks post intervention)
  Depression measured using the Beck Depression Inventory (range score from 0 [better status] to 63 [severe depression])
Fear Avoidance Beliefs | Baseline; 8 weeks measurement (post intervention); 32 weeks measurement (24 weeks post intervention)
  Fear Avoidance Beliefs measured using the Fear Avoidance Belief Questionnaire (range score from 0 [Lower levels of fear-avoidance beliefs] to 96 [higher levels of fear-avoidace beliefs])
Fear Avoidance Components | Baseline; 8 weeks measurement (post intervention); 32 weeks measurement (24 weeks post intervention)
  Fear Avoidance Beliefs measured using the Fear Avoidance Components Scale (range score from 0 [Lower levels of fear-avoidance components] to 100 [higher levels of fear-avoidace components])
Adherence | Baseline; 8 weeks measurement (post intervention); 32 weeks measurement (24 weeks post intervention)
  Adherence measured using the TRAK application
Adherence | Baseline; 8 weeks measurement (post intervention); 32 weeks measurement (24 weeks post intervention)
  Adherence measured using an exercise diary

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo Martín-San Agustín, PhD, Principal Investigator — University of Valencia
Locations (1):
- University of Valencia, Valencia, Select One, Spain

IPD SHARING:
Plan to Share IPD: No